

# Part 1: Subject Information Sheet (SIS)

| Sub | ject | ID | (6 | dig | gits | ): |
|-----|------|----|----|-----|------|----|

Short title: A Phase IIb study on influenza Vaccine Candidate (FLU-v)

Protocol Title: A randomised, double-blind, placebo-controlled, single-centre phase IIb trial as part of the EU-funded UNISEC project to assess the immunogenicity and safety of different formulations and dosing regimens of FLU-v vaccine administered subcutaneously in healthy adults aged 18-60 years.

**Sponsor: SEEK** 

Protocol Version: 4.0 Dated 17 June 2016

Sponsor Code: FLU-v 003

**EudraCT Number: 2015-001932-38** 

NL55061.000.15

#### Dear Sir / Madam

You are being asked to participate in a research study. Before you decide it is important for you to understand why the research is being done and what it will involve. Please take time to read the following information carefully and the general brochure: 'Medisch Wetenschappelijk Onderzoek' (Medicinal Research Involving Human Subjects) appendix 4. Ask us if there is anything that is not clear or if you would like more information. Take time to decide whether or not you wish to take part.

## 1. Background to the study

The Influenza virus is one of the major known viruses passed from person to person and these viruses are changing constantly. Due to these virus changes there are new flu strains appearing and the traditional flu vaccine preparation can't always accurately predict these changes on time to prepare an effective vaccine and when it fails people can get infected even if vaccinated.

The pharmaceutical company SEEK [known as the Sponsor] has a new flu vaccine, the "test vaccine", called **FLU-v** and it is currently under investigation and is not yet available to the general public. FLU-v is a vaccine that aims to protect against all strains of flu (universal vaccine) and therefore eliminates the need to develop a new vaccine every year. The sponsor is a member of the Universal Flu Vaccines Secured (UNISEC) consortium, experts in flu vaccine research and development. The consortium conducts research to find out which flu vaccines can successfully combat existing flu viruses, any new emergent flu viruses and also to be able to get approval to vaccinate worldwide. This consortium is funded by the European Union. The **FLU-v 003** vaccine study will play an important role in this research and development between the UNISEC group and SEEK, which will be clinically tested in partnership with the Isala Hospital in Zwolle [known as the study centre].



#### 2. What is the purpose of this study?

The purpose of this study is to see what effect **FLU-v** will have on your body in fighting against multiple types of flu viruses. This study will look at how safe FLU-v is when administered, how it is tolerated in your body and to see how successful it is in preventing flu or reducing the severity of the flu symptoms

You will be in this study for a maximum of 7 months. 222 subjects will take part in this study, which will be conducted at Isala Hospital in Zwolle.

# 3. Do I have to take part?

Taking part in the study is entirely voluntary. It is up to you to decide whether or not to take part in the study. If you decide to take part, you will be given this Subject Information Sheet (SIS) to keep and be asked to sign an Informed Consent Form (ICF). Once you are in the study you are still free to withdraw at any time and without giving a reason, you must however inform your study doctor and return to the study centre for a final check-up.

# 4. What does this study mean for me?

If you agree to take part in the study, the study doctors will examine you to make sure you are eligible to enter the study. The initial examination will consist of testing a 15ml sample of your blood (a tablespoon) to check general health, measure antibodies of the flu in your blood, physical exam (weight, blood pressure and heart rate), medical history/medications taking (prescription and non-prescription)and personal information (ethnic origin, gender and date of birth). You will not be able to take part in this study if you have received the traditional flu vaccine in the past 6 months. For more information regarding this initial visit please refer to **appendix 3**.

If you are female and of childbearing age, you must agree to use effective contraceptive methods, such as hormonal contraceptive plus a barrier contraceptive. A blood pregnancy test will be performed at your first study visit. If you are pregnant or breast feeding, you will not be allowed to take part in the study. Males must agree to practice appropriate contraception whilst taking part in the study also.

If you are found to be eligible, you may enter the study. You will be asked to sign and date the informed consent form before proceeding further.

At the next study visit you will be randomly allocated to **one** of the four treatment groups summarised below;

- Treatment 1: FLU-v (test vaccine) injection at the study start (Day 0) and then again 21 days later
- ➤ Treatment 2: FLU-v (test vaccine) with an additional substance added [known as ISA 51] which improves the effect of the test vaccine. Injection will be given at the study start (Day 0) and then Placebo (no test vaccine) alone 21 days later
- Treatment 3: Placebo (no test vaccine) injection on both the study start (Day 0) and then 21 days later
- > Treatment 4: Placebo (no test vaccine) with an additional substance added [known as ISA 51] at the study start (Day 0) and then Placebo (no test vaccine) alone 21 days later

#### > Randomisation

You will be placed into one of the four treatment groups. For this division to be carried out as scientifically as possible each study subject will be randomly (like the flip of a coin) assigned to one



of four treatment groups. This process is referred to as randomisation. Your study doctor will have no influence on the result of the randomisation.

For every three subjects taking part in the study, two will receive the test vaccine and one will not. Half of the people receiving the test vaccine will receive two doses and the other half will receive just one dose of the test vaccine.

# > Double Blind Study

➤ Neither you nor the study team will know which treatment you are randomised to receive. This information will be kept confidential unless required. This is called a double blind study. By comparing the 4 treatment groups it can then be seen if one treatment is more effective than another and whether it has more or less side effects.

Every subject in the study will receive a total of 2 injections just under the skin of the upper non-dominant arm, one at the start and the second 21 days later. The treatment group you are randomised to (1-4), will determine what you will receive.

You will be required to attend a total of 5 subject visits. **Appendix 1** shows you a detailed overview of the study procedures and visits.

Once enrolled on the study you will be asked to give a further 3 blood samples, approximately 60mls (4 tablespoons) at the beginning of the study (Day 0), Day 42 and Day 180 - in total, approximately 180ml of blood (12 tablespoons) will be collected over the three visits.

You will also be asked to complete a diary card to write down any side effects that you may experience after you have been given the study injection. You should take this diary card along with you to each of your study visits where the study doctor will discuss this with you.

After the 3<sup>rd</sup> visit to the study centre you will be given an additional diary card to document any subsequent flu-like symptoms you may experience. These diary cards will need to be completed daily until the study has concluded. Additionally, we would ask you to also call the study centre if you experience flu-like symptoms to arrange the collection of a nose and tonsil swab to confirm whether you have the flu or not.

Biological samples (i.e. blood samples, nasal and tonsil swabs) will be used only for this study and be transported to central laboratories outside the Netherlands for UNISEC project immune response testing. The samples will be destroyed after 10 years from the study completion. Transferring biological samples from one country to another is performed according to approved and applied European legislation.

The study period is a maximum of 7 months. However, your participation may cease earlier if:

- (1) You do not follow the study requirements,
- (2) You wish to stop the study of your own free will,
- (3) If the study staff, the independent ethics committee (IEC)/ independent regulatory board (IRB) or the Sponsor (SEEK) consider it desirable to stop your participation. This will be discussed with you,
- (4) Or if new information is found which after careful review, the study staff, independent ethics committee/independent regulatory board or the Sponsor feel that it is in your best interests to no longer be in the study.



#### 5. What are the alternatives for treatment?

There are other flu vaccines approved for use. Your study doctor will be able to explain these other vaccination possibilities should you wish to find out. However, they will not be provided as part of this study as this is a specific controlled clinical study to determine if the **FLU-v** vaccine is effective against the flu virus

You can't take part in the study if you have been vaccinated with any other influenza vaccine in the last 6 months.

# 6. What are the possible advantages and disadvantages/risks in participating in this study?

The **FLU-v** vaccine is aiming to protect against a broad range of flu types, however the vaccine is still under research. Since the **FLU-v** vaccine is still a test vaccine you may not receive any direct medical benefits from taking part in the study. In addition, there is also a chance of you just receiving a placebo (no test vaccine).

Once enrolled in the study you will be required to attend for a total of 5 visits for study procedures and to keep track and report side effects/ FLU-like symptoms to the study staff, if you experience them. If you do experience flu-like symptoms you will be required to attend an extra visit to collect a nasal/tonsil swab. In addition, in the unlikely event that you feel unwell during the course of the study, the study doctor may ask you to attend an additional visit to monitor your symptoms. For a more detailed description of study procedures and visits, please see **appendix 1**.

It is possible that if the test vaccine was given to a pregnant woman this may harm the unborn child. Pregnant women are therefore excluded from taking part in this study. Women who are at risk of becoming pregnant will be asked to have a pregnancy test before taking part to exclude the possibility of an unknown pregnancy. Effective contraception must be used for both males and females for the duration of the study and your study doctor will discuss this with you. Any woman who finds that she has become pregnant while taking part in the study should immediately tell the study doctor.

#### 7. What side effects can you expect?

All medications can cause side effects, although not everybody gets them. Possible known side effects associated with the **test** vaccine are;

Redness, swelling, pain and / or itching at the site of injection, fever / temperature, chills, headache, nausea, fatigue, myalgia and mild flu-like symptoms may occur. There may also be changes in some of your blood values, but these are usually mild and not significant.

These side effects are usually more common at the start of the study and typically don't last more than a few days. You may experience side effects that are not yet known and this is the reason why you will be asked to complete a study diary card of all symptoms you may be experiencing and bring with you when you attend the study centre.

## 8. What happens if you no longer wish to take part?

Your participation is entirely voluntary and you can decide at any point during the course of the study whether to take part or not. If you decide not to take part, you do not need to do anything. You do not have to sign anything. You do not have to give a reason for not participating or withdrawing your consent.



#### 9. What happens if new information becomes available?

Sometimes during the course of a study, new information on the vaccine that is being investigated becomes available. Should this occur, your study doctor or nurse will inform you and discuss further whether you want to proceed with the study or not. If you do decide to continue to take part in the study, you will be asked to sign an updated consent form which will contain any new information and will be approved by the ethics committee. Alternatively, the study doctor may also decide that it is in your best interests to withdraw you from the study. Your study doctor will explain the reasons for this and will make sure that you continue to receive the best care.

# 10. What happens when the study has completed?

The study will last for a maximum of about 7 months from the time you sign the consent until study conclusion. Your participation may end earlier for many reasons as previously discussed. No further medical care is anticipated after study completion.

#### 11. Are you insured when you take part in the study?

For everyone who participates in this study an insurance policy is taken out. The insurance covers damage resulting from participation in the study which would not have occurred if you did not participate in this study. **Appendix 2** provides more information about the insurance.

## 12. Usage and storage of your data and biological samples

For this study it is necessary to collect and use biological samples (Blood and Nasal/Throat swabs) and your medical and personal data. You will receive a code that will be marked on your data and the biological samples. Your name and personal identifiers will be deleted.

## Your data:

Medical and personal data collected for this study on you includes;

➤ General health data, physical exam (weight, blood pressure and heart rate), medical history/medications taking (prescription and non-prescription) and personal information (ethnic origin, gender and date of birth)

This data will remain confidential. The investigators at the hospital are the only people who know which code you have.

You may cancel your permission for the investigators to collect any new medical and personal data for the study. This can be done at any time during the study by contacting your study doctor. If you cancel your permission, you will not be able to stay in the study. The study staff will stop collecting any new medical and personal data about you. All your medical and personal data collected up to that point will used for analyses.

We will share the medical and personal data with the sponsor of the study but only using the code and never using your name. The key to the code will stay with the investigator. In the reports/publications about the study only the code will be used.



Some people may have access to your medical and personal data. This is to check that the study is done properly. General information about this can be found in the general brochure on medical research (appendix 4).

People who may access your data are:

- the study team
- the manufacturer of FLU-v vaccine
- a monitor who has been commissioned by the Sponsor
- the Healthcare Inspectorate (IGZ) and MHRA.

They will keep your medical and personal data a secret. If you sign the consent form, you consent to your medical and personal data being collected, stored and accessed.

All your medical and personal data will be protected in accordance with the European data protection legislation. Your medical and personal coded data, including sensitive data, will be transferred to the Sponsor (SEEK) and their representatives and to regulatory authorities both within and outside the European Union (EU). By signing this consent form you are giving permission for this to happen.

The investigator will store your data for 15 years

The sponsor of the study will receive a copy of the medical and personal coded data without your name and will store the data for 15 years as well.

## Your Biological Samples (Blood samples and Nasal/Tonsil Swabs):

Your biological samples collected during the course of the study will be sent to the following centres for the analyses of your immune response:

- Norwegian Institute of Public Health. Norway
- Robert Koch Institute. Germany

The European guidelines for personal data protection do apply here and your biological samples will be sent in encoded form (no name or personal identifiers).

We will keep your biological samples for 10 years. We may need to use them for additional research in the future. It will still concern research on immune responses to the test vaccine. You can indicate whether you agree with this on the consent form. You can always withdraw consent at anytime and your biological samples will then be destroyed. If your samples have already been analysed the results will be used.

This study is listed in a clinical trial registry called **ClinicalTrials.gov**. The website does not contain any information that can identify you. The website may contain a summary of the study results once the study is completed. You may find the study under FLU-v 003 (EudraCT number: 2015-001932-38).

General information about the registration of research can be found in the general brochure on medical research (appendix 4).

# 13. What happens with the results of the study?

The results of the study will be analysed and may be published in scientific and medical journals. The data may also be used to support the registration and marketing of the test vaccine. The unique coding will ensure that you are not identifiable any report or publication.

# 14. Are there any extra costs/ will compensation be provided if you decide to participate in the study?



There are no costs for you to pay if you wish to participate in the study. The study treatment will be provided free of charge by the Sponsor of the study. The study Sponsor will also be responsible for all procedures that are solely performed for the purpose of this study. The study doctor at Isala Hospital will be paid by the Sponsor for your participation in the study. You will not be charged for your study test vaccines, visits to your study doctor, study-related exams, tests, or procedures. The travel expenses you incur whilst participating in this study will be reimbursed up to €15.00.

#### 15. Who has reviewed and approved the study?

The Central Committee on Research involving Human Subjects (CCMO) has approved the study. Approval means that the commission is convinced that your rights are respected, any risks are minimized and weighed against the potential benefits, and that you are given enough information to make an informed decision to take part in the study.

#### 16. Who will be informed of my study participation?

To ensure your safety and ongoing medical care we will liaise with your primary care physician about your study participation.

Your primary care physician may give in confidence details of your relevant medical or drug history. Results of any assessment or medical history obtained during the course of this study may be shared with your primary care physician. You need to give permission for this on the consent form at your initial visit.

# 17. Do you need additional study information?

If you have any questions before or at any point during the course of the study, please contact the study doctor or the study nurse.

The study contact details are as follows:

Study Doctor: Dr. Paul Groeneveld, Dr. Deenweg 2, 8025 AB Zwolle, TEL: 038 4243350 (secr. Interne Geneeskunde)

The study nurse Lonneke Buitenhuis, TEL 038-424-8221.

# 18. Study Concerns or Complaints

If you have any concerns during the study, please contact the independent doctor who is not involved in the study but who is an expert in the area of this research. Prof. Dr. P.L.P. Brand has been appointed as the study independent doctor. You may also contact the independent doctor if you have questions that you would prefer not to discuss with the study doctor before or during the study.

- Independent doctor: Prof. Dr. P.L.P. Brand, TEL: 038-4245050 Email: p.l.p.brand@isala.nl

If you have any comments, complaints or problems, then discuss them as possible with the nurse, study doctor or independent doctor. If you do not find desirable a conversation with them or are dissatisfied with the proposed solution, please contact the complaints officer. The complaints officer will listen to your complaints, assisting as necessary in the draft script of your complaint and mediate between you and the person about whom you are complaining. Also, it shall inform you of the complaints and the procedure for liability. If your complaint is not resolved to your satisfaction, or if you do not want to not contact the complaints officer, you can file a written complaint.



You can contact the complaints officer through the secretariat Complaints Care, (038) 424 47 27, Monday through Friday, available from 9:00 to 15:00 pm.

Mailing address:

Isala

Complaints Reception, Attn: Complaints Officer

PO Box 10400

8000 GK Zwolle

You can also submit a complain online via the following website: http://www.isala.nl/patienten/rechten-plichten-en-klachtenbehandeling/klachtenbehandeling

# 19. Appendix

- 1. Detailed Description of study visits and procedures
- 2. Insurance policy
- 3. Blood sample screening visit
- 4. General Brochure Medicinal Research Involving Human Subjects



# Part 2: Informed Consent Form (ICF)

| Subject I | D (6 | digits | ): |
|-----------|------|--------|----|

Protocol Title: A randomised, double-blind, placebo-controlled, single-centre phase IIb trial as part of the EU-funded UNISEC project to assess the immunogenicity and safety of different formulations and dosing regimens of FLU-v vaccine administered subcutaneously in healthy adults aged 18-60 years.

Short Title: A Phase IIb study on influenza Vaccine Candidate (FLU-v)

Protocol Version: 4.0 Dated 17 June 2016

Sponsor Code: FLU-v 003

EudraCT Number: 2015-001932-38

NL55061.000.15

Name of Investigator: Dr Paul Groeneveld

| | Your consent | Please initial box |
|---|---|---|
| 1. | I confirm I have read and understood the <b>subject information sheet</b> dated (* <b>insert date</b> ) version(* <b>insert version number</b> ) for the above study and have had time to consider the information. I have had a chance to ask questions and have had these questions answered to my satisfaction. | |
| 2. | I agree to my primary care physician being informed that I am taking part in this study. I agree that my primary care physician can give in confidence details of my relevant medical or drug history to Isala Hospital. I agree that the Investigator can send any health results or medical history obtained during this study to my primary care physician. | |
| 3. | I confirm that I understand and agree to abide by the restrictions and birth control advice. If you are female and of childbearing age, you must agree to use effective contraceptive methods, such as hormonal contraceptive plus a barrier contraceptive. Males must agree to practice appropriate contraception whilst taking part in the study. | |
| 4. | I understand that agreeing to take part in this study is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | |
| 5. | I consent to give 15 ml blood for the screening blood tests and measuring antibodies against the flu. | |
| 6. | I understand that if I do not meet the inclusion/exclusion criteria or the test results show any abnormal value or a positive pregnancy (females), I will not be able to participate in the study. | |



| 7. | I understand that in addition to the pre-study (screening) blood<br>need to give blood samples for immune response follow-up. 60<br>taken on day 0, 42 and 180. A total of 180 ml blood will be take<br>sampling times. | ml will be |
|---|---|---|
| 8. | I understand that I need to contact Isala Hospital immediately if I influenza like illness during the influenza season (1st December April 2017). The nasal and tonsil swabs will be taken within 4 day start of the symptoms. | 2016 to 1 <sup>st</sup> |
| 9. | I understand that biological samples (i.e. blood samples, nass swabs) will be used only for this study and be transported laboratories outside the Netherlands for UNISEC project immune testing. The samples will be destroyed after 10 years from completion. You can always withdraw consent at anytime biological samples will then be destroyed. If your samples had been analysed the results will be used. Transferring biological samples one country to another will be performed according to approved a European legislation. | to central e response the study and your ve already mples from |
| 10. | I understand that relevant sections of my medical notes and collected during the study may be looked at by the Sponso appointed representatives (monitors and auditors), study investigated in the study investigated in the study investigated in the study. I give permission for these individuals to have access to mean to my taking study. I give permission for these individuals to have access to mean taking in the study. | r's (SEEK)<br>stigators at<br>RA) or the<br>part in this |
| 11. | I agree to the transfer of my medical and personal coded data sensitive data, to the Sponsor (SEEK) or their representative regulatory authorities both within and outside the European Unit agree that my personnel coded data may be archived. | res and to |
| 12. | I understand that my study coded research data will be kept for after the study completion. Data will be permanently removed computer network afterwards. | - |
| 13. | I agree to take part in the above study and will be given a sign copy of the Subject Information Sheets (SIS) and Informed Cor (ICF). | |
| Name of Subject | Date (DD/MMM/YYYY) Signatur | re |
| Name of the personal Taking the conser | , | re |



# Appendix 1. Detailed description study procedures and visits

#### **Procedures**

You will receive two vaccinations with an interval of 21 days (day 0 and 21). On both occasions you will receive one injection with 0.5 milliliter of the vaccine (500 micrograms FLU-v) or placebo, alone or with the adjuvant (ISA 51) underneath the skin in your upper arm. It is planned that 222 subjects (men and women aged between 18 and 60 years) will participate in the study. You will be allocated by random (flipping a coin) to one of the four treatment groups – you will not have a choice to which group you are allocated;

| Group | Treatment | Number of Subjects | |
|---|---|---|---|
| Croup | Day 0 | Day 21 | Training of Gangoote |
| 1 | Vaccine | Vaccine | 74 |
| 2 | Vaccine plus adjuvant | Placebo | 74 |
| 3 | Placebo | Placebo | 37 |
| 4 | Placebo plus adjuvant | Placebo | 37 |

# Screening (Visit 1)

The screening visit includes one visit to your site with the purpose of checking if you can participate in the study. You can participate in the study if you don't have any medical conditions, a negative pregnancy test (females) or medicines that could affect your safety when taking part in the study or influence the results obtained during the study.

After the study has been explained to you and you are happy that all your questions have been answered you will be asked to sign the consent form. The study staff will then ask several questions about your alcohol, drugs and cigarette consumption, ethnic group, gender, age, medical history and medications and flu shots you have had recently. In addition, the study doctor will perform a physical examination which contains measuring blood pressure, heart rate, respiration, temperature, height and weight. You will also be asked to give blood samples for laboratory tests and a pregnancy test (females). These blood tests are performed as a general health check and also to ensure that you do not have an increased risk of adverse reactions to this vaccine.

#### First dose - Day 0 (Visit 2)

You will be examined by the study doctor. If your temperature is higher than 38 degrees Celsius, you will not be able to proceed with the study. We will take approximately 60 ml of blood from one of the veins in your arm to measure the immune response of your body before the vaccine is administered for the first time. The vaccine will be given in your upper arm. The vaccine is designed to be administered with a needle and is placed just beneath the skin. This may cause some mild discomfort during the injection.



For your safety, we would ask you to please remain for at least 30 minutes in the clinic after the injection for observation for any immediate side effects from the injection.

You will receive; an Adverse Event Diary Report Card to keep track of any side effects that may occur until the 3<sup>rd</sup> visit on Day 42 visit and a thermometer to check your temperature. You will be instructed about what you should include in the diary, and you will be instructed how to measure skin reactions and temperature.

## Second dose - Day 21 (Visit 3)

You will be asked to return to the clinic. Your Adverse Event Diary Report Card of side effects will be collected from you and assessed. You will be examined by the study doctor. If your temperature is above 38 degrees Celsius at this visit, you cannot proceed with the study. The vaccine will be given in your upper arm as per the previous visit.

#### Check - Day 42 (Visit 4)

You will be asked to return to the clinic where 60 ml of blood is collected. The visit lasts approximately one hour

You will be given a Flu Symptom Diary Card which needs to be completed daily during the influenza season (1<sup>st</sup> December 2016 to the 1<sup>st</sup> April 2017). The study nurse will explain each symptom listed on the card and how to complete it.

# Last visit clinic - Day 180 (Visit 5)

You will be asked to return to the clinic where 60 ml of blood is collected. The visit takes about 1 hour.

#### From Visit 5 visit to the end of the study

You will complete daily the Symptom Diary card and mail/fax/email them to the clinic every two weeks. Also you will be asked to contact the clinic if you feel unwell for 24 hours with a sudden onset of at least:

- One respiratory (cough, sore throat, shortness of breath, runny nose, stuffy nose, sneezing or earache) and
- One systemic symptom (fever, malaise, headache and myalgia (muscle and joint pain)).

The study nurse will decide based on your symptoms if it is necessary to collect a nose and throat swab to confirm whether you have the flu or not.

We will ask you to contact the clinic if you experience any side effects that you wish to discuss or seek advice on.



## **Appendix 2: Insurance**

For anyone who takes part in this research, SEEK (The Sponsor) has taken out insurance. The insurance covers damage caused by participation in the research. This applies to damage during the trial or within four years after its end. Damage must be reported to the insurer within four years. The insurance does not cover all damage. Below this text you find a short description about the damage which is not covered by insurance.

These provisions are contained in the Decree on compulsory insurance for medical research involving humans. This decision can be found on the website <a href="www.ccmo.nl">www.ccmo.nl</a>, the website of the Central Committee on Research involving Human Subjects (see "Library" and then "Laws"). In case of damage you can make direct contact with the insurer.

# The insurer of the study is: **Chubb Insurance Company**

The insurance provides coverage of € 650,000 per participant, € 5 million for the entire research and € 7,5 million per year for all investigations conducted by the same client).

The insurance does **not** cover the following damage:

- damage due to a risk where you have been informed with in the written information. This does not apply if the risk was more severe than was anticipated or if the risk was very unlikely;
- damage to your health that would also have occurred if you had not participated in the study;
- damage due to not (completely) following the directions or instructions;
- damage to your offspring, as a consequence of a negative effect of the study on you or your offspring;
- damage from an existing treatment method in research on existing treatments



#### Appendix 3: Blood sample screening visit

At the screening visit, a blood sample is taken to check your general health. Routine blood tests will be performed to make sure that you have no increased risk of side effects of the vaccine. Laboratory tests will be carried out in order to examine the blood (hematology and serum chemistry) and a pregnancy test for females. Blood levels should be within the normal range and pregnancy test should be negative. Blood levels outside the normal range are only acceptable for the study after the investigator has determined that the abnormal values are not "clinically significant".

If you have any abnormal test results or a positive pregnancy test, you cannot participate in the study. We recommend that you then contact your primary care physician for further investigation or come along to the Isala Hospital for a consultation.

In addition to the routine blood test, serum of the collected blood will be used for testing before you start the study to see if you already have protective responses to the flu viruses present during the upcoming influenza season (1<sup>st</sup> December 2016 to 31<sup>st</sup> March 2017).

Blood samples will be used only for this study and will be retained as long as the quality of the samples are not affected and the samples will be kept for no longer than 10 years after the end of the study.